CLINICAL TRIAL: NCT00631462
Title: A Phase 1, Open-label, Dose-escalation Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Orally Administered TG101348 in Patients With Primary, Post-polycythemia Vera, or Post-essential Thrombocythemia Myelofibrosis
Brief Title: A Dose-escalation Study of the Safety and Tolerability of Orally Administered TG101348 in Patients With Myelofibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TargeGen (Industry)
Responsible Party: Jolene Shorr, TargeGen, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MF-TG101348-001
Record Dates: First submitted 2008-01-29; First posted 2008-03-07 (Estimated); Last update posted 2009-10-26 (Estimated); Status verified 2009-10

CONDITIONS: Myelofibrosis
Keywords: primary myelofibrosis; post-polycythemia vera myelofibrosis; post-essential thrombocythemia myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — fedratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: TG101348

INTERVENTIONS:
Drug: TG101348 — Orally administered, once a day, for 28 days, up to 6 cycles.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of orally administered TG101348 in patients with myelofibrosis.

DETAILED DESCRIPTION:
TG101348 is a potent small molecule inhibitor of Janus kinase 2 (JAK2). This is a first-in-human study that will include a dose-escalation phase, to establish the maximum tolerated dose, and an expanded cohort, dose-confirmation phase. The safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary clinical activity of TG101348 in patients with myelofibrosis will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myelofibrosis (primary, post-polycythemia vera, or post-essential thrombocythemia)
* At least 18 years of age.
* ECOG PS 0, 1, or 2.

Exclusion Criteria:

* Any chemotherapy, immunomodulatory therapy, immunosuppressive therapy, corticosteroids, or growth factor treatment within 14 days prior to initiation of study drug.
* Major surgery or radiation therapy within 28 days prior to initiation of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Safety (i.e., adverse events; effects on laboratory parameters, vital signs, and ECGs; dose-limiting toxicities), tolerability, and MTD | 28 days

SECONDARY OUTCOMES:
Pharmacokinetics and pharmacodynamics | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Ayalew Tefferi, MD, Study Chair — Mayo Clinic
Locations (6):
- United States (6):
  - UCSD Moores Cancer Center, San Diego, California
  - Stanford Comprehensive Cancer Center, Stanford, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MPD Foundation — http://mpdfoundation.org/